CLINICAL TRIAL: NCT06015698
Title: Laparoscopic Tubal Disconnection Versus Laparoscopic Salpingectomy in Infertile Patients Scheduled for IVF/ICSI. Randomized Controlled Trial
Brief Title: Laparoscopic Tubal Disconnection Versus Laparoscopic Salpingectomy in Infertile Patients
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Ain Shams Maternity Hospital (Other)
Responsible Party: Principal Investigator, Ahmed Mohammed Elmaraghy, Lecturer in Obstetrics and Gynecology, Ain Shams Maternity Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 10
Record Dates: First submitted 2023-08-23; First posted 2023-08-29 (Actual); Last update posted 2023-08-29 (Actual); Status verified 2023-08

CONDITIONS: Infertility, Female
MeSH Terms: conditions — Infertility, Female

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Tubal disconnection (Experimental): 1. The tube is grasped in the isthmic portion of the tube at least 2cm from the cornua. Bipolar coagulation will provide a more localized area of tubal burn so requiring at least 3cm of the tube to be coagulated
  2. The electrosurgical generator should set to deliver a power of 25W in nonmodulated mode to desiccate tissue sufficiently
  3. The tube should be coagulated with 2 to 3 contiguous burns to provide an area of about 3cm of coagulation. Th endpoint of coagulation is cessation of the current flow
  4. Then, the tube is severed in the middle of the burn area with laparoscopic scissors
  5. Ensure adequate hemostasis
  Interventions: Procedure: Laparoscopic tubal disconnection
- Salpingectomy (Active Comparator): 1. The tube will be removed from its anatomical attachements by progressive bipolar coagulation
  2. Progressive coagulation and cutting of the mesosalpinx begins at the proximal isthmus of the tube and progresses to the fimbriated end using bipolar coagulation and laparoscopic scissors
  3. Removal of the tube through one of the ancillary ports using artery forceps
  4. Ensure adequate hemostasis
  Interventions: Procedure: Laparoscopic salpingectomy

INTERVENTIONS:
Procedure: Laparoscopic tubal disconnection — 1. The tube is grasped in the isthmic portion of the tube at least 2cm from the cornua. Bipolar coagulation will provide a more localized area of tubal burn so requiring at least 3cm of the tube to be coagulated
  2. The electrosurgical generator should set to deliver a power of 25W in nonmodulated mode to desiccate tissue sufficiently
  3. The tube should be coagulated with 2 to 3 contiguous burns to provide an area of about 3cm of coagulation. Th endpoint of coagulation is cessation of the current flow
  4. Then, the tube is severed in the middle of the burn area with laparoscopic scissors
  5. Ensure adequate hemostasis
  Arms: Tubal disconnection
Procedure: Laparoscopic salpingectomy — 1. The tube will be removed from its anatomical attachements by progressive bipolar coagulation
  2. Progressive coagulation and cutting of the mesosalpinx begins at the proximal isthmus of the tube and progresses to the fimbriated end using bipolar coagulation and laparoscopic scissors
  3. Removal of the tube through one of the ancillary ports using artery forceps
  4. Ensure adequate hemostasis
  Arms: Salpingectomy

SUMMARY:
Tubal factor infertility is known to be one of the most common indications for IVF treatment. Patients with hydrosalpinges have been identified to have poor pregnancy outcomes such as lower implantation and pregnancy rates & higher rates of spontaneous abortion and ectopic pregnancies. Surgical intervention can be recommended for patients with hydrosalpinx prior to IVF/ICSI.

This study will be done at Ain Shams University Maternity Hospital, to compare laparoscopic salpingectomy & laparoscopic tubal disconnection as two surgical modalities of treatment of unilateral or bilateral hydrosalpinges in women older than 30 years and scheduled for IVF/ICSI, regarding implantation rates, clinical pregnancy rates, ongoing pregnancy rates, ectopic pregnancy rates, and operative complications.

DETAILED DESCRIPTION:
It is estimated that tubal factors account for 14% of the causes of subfertility in women. The prevalence of hydrosalpinx among tubal diseases is as high as 30% of couples presenting with infertility from tubal factors.

Hydrosalpinx is the dilation of the fallopian tube in the presence of distal tubal occlusion, which may result from several causes. The leading cause of distal tubal occlusion is pelvic inflammatory disease (PID), usually resulting from a prior sexually transmitted disease, such as Chlamydia trachomatis or Neisseria gonorrhoeae. Tubal tuberculosis is an uncommon cause of hydrosalpinx, though re-emerging in developed countries. Other etiologies include endometriosis, appendicitis, and abdominopelvic surgery.

Depending on several patient factors, tubal microsurgery, or more commonly IVF with its improving success rates, are the recommended treatment options for tubal factor infertility.

In addition to its essential role in infertility, hydrosalpinx has an adverse effect on the outcome of in vitro fertilization (IVF) Hydrosalpinx can decrease the clinical pregnancy rate of IVF-ET, and increase the incidence of abortion and ectopic pregnancy.

The presence of hydrosalpinx has a negative effect on IVF/ET because of the suspected embryotoxicity of the hydrosalpingeal fluid due to a combination of mechanical and chemical factors thought to disrupt the endometrial environment.

Surgical treatment should be considered for all women with hydrosalpinges prior to IVF treatment (Johnson et al .,2004 )

Removing (salpingectomy) or occluding blocked or diseased fallopian tubes before IVF can increase pregnancy and live birth rates for women on the IVF program.

A network meta-analysis showed that Proximal tubal occlusion, salpingectomy, and aspiration for treatment of hydrosalpinx scored consistently better than did no intervention for the outcome of IVF/ET. Tubal occlusion and salpingectomy also improve ongoing pregnancy rates. Proximal tubal occlusion ranks highest for most of the outcomes assessed, whereas no intervention scores consistently as the least effective strategy for all outcomes

ELIGIBILITY:
Inclusion Criteria:

1. Infertile ( primary or secondary ).
2. Age > 30 years .
3. HSG with unilateral or bilateral hydrosaalpinx , confirmed laparoscopically.
4. Scheduled for IVF/ICSI

Exclusion Criteria:

1. Contraindications for laparoscopy

   * Cardiac disease.
   * BMI > 40 kg/m²
   * Previous midline incision .
   * Past history of TB peritonitis .
2. Proximal tubal block by HCG .
3. Frozen pelvis proved by previous laparoscopy or laparotomy .
4. Allergy to contrast media of HSG .
5. Premature ovarian failure (Serum FSH >40 mIU/ml )
6. Prescence of Male factor contributing to the infertility proved by abnormal semen analysis
7. Prescence of Ovarian factor contributing to the infertility proved by the prescence of features suggesting anovulation

Ages: 30 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 150 (Estimated)
Dates: Start 2023-08-30 (Estimated); Primary Completion 2024-08-30 (Estimated); Study Completion 2024-08-30 (Estimated)

PRIMARY OUTCOMES:
Ongoing pregnancy rate | From 10 + 0 weeks of gestation
  Pregnancy with detectable heart beat 10weeks gestation or beyond

SECONDARY OUTCOMES:
Operative time | in minutes starting from laparoscopic entry into the peritoneal cavity till removal of the primary trocar from the cavity
  in minutes starting from laparoscopic entry into the peritoneal cavity till removal of the primary trocar from the cavity
Intraoperative complications | During the procedure
  Bowel injury - Vascular injury
Postoperative complications | First 48 hours after the procedure
  ileus - surgical emphysema

CONTACTS AND LOCATIONS:
Overall Officials: Hamdy B Alqenawy, M.D.,, Study Director — Ain Shams university - Faculty of Medicine; Ahmed G Abd Elrahim, M.D.,, Principal Investigator — Ain Shams university - Faculty of Medicine; Alaa S Elsewafy, M.D.,, Principal Investigator — Ain Shams university - Faculty of Medicine

REFERENCES:
- [Background] Ajonuma LC, Ng EH, Chan HC. New insights into the mechanisms underlying hydrosalpinx fluid formation and its adverse effect on IVF outcome. Hum Reprod Update. 2002 May-Jun;8(3):255-64. doi: 10.1093/humupd/8.3.255. PMID 12078836
- [Background] D'Arpe S, Franceschetti S, Caccetta J, Pietrangeli D, Muzii L, Panici PB. Management of hydrosalpinx before IVF: a literature review. J Obstet Gynaecol. 2015;35(6):547-50. doi: 10.3109/01443615.2014.985768. Epub 2014 Dec 1. PMID 25436898
- [Background] Dreyer K, Lier MC, Emanuel MH, Twisk JW, Mol BW, Schats R, Hompes PG, Mijatovic V. Hysteroscopic proximal tubal occlusion versus laparoscopic salpingectomy as a treatment for hydrosalpinges prior to IVF or ICSI: an RCT. Hum Reprod. 2016 Sep;31(9):2005-16. doi: 10.1093/humrep/dew050. Epub 2016 May 21. PMID 27209341
- [Background] Dun EC, Nezhat CH. Tubal factor infertility: diagnosis and management in the era of assisted reproductive technology. Obstet Gynecol Clin North Am. 2012 Dec;39(4):551-66. doi: 10.1016/j.ogc.2012.09.006. PMID 23182560
- [Background] Hong X, Ding WB, Yuan RF, Ding JY, Jin J. Effect of interventional embolization treatment for hydrosalpinx on the outcome of in vitro fertilization and embryo transfer. Medicine (Baltimore). 2018 Nov;97(48):e13143. doi: 10.1097/MD.0000000000013143. PMID 30508891
- [Background] Johnson N, van Voorst S, Sowter MC, Strandell A, Mol BW. Surgical treatment for tubal disease in women due to undergo in vitro fertilisation. Cochrane Database Syst Rev. 2010 Jan 20;2010(1):CD002125. doi: 10.1002/14651858.CD002125.pub3. PMID 20091531
- [Background] Nackley AC, Muasher SJ. The significance of hydrosalpinx in in vitro fertilization. Fertil Steril. 1998 Mar;69(3):373-84. doi: 10.1016/s0015-0282(97)00484-6. PMID 9531862
- [Background] National Collaborating Centre for Women's and Children's Health (UK). Fertility: Assessment and Treatment for People with Fertility Problems. London: Royal College of Obstetricians & Gynaecologists; 2013 Feb. Available from http://www.ncbi.nlm.nih.gov/books/NBK247932/ PMID 25340218
- [Background] Ng KYB, Cheong Y. Hydrosalpinx - Salpingostomy, salpingectomy or tubal occlusion. Best Pract Res Clin Obstet Gynaecol. 2019 Aug;59:41-47. doi: 10.1016/j.bpobgyn.2019.01.011. Epub 2019 Jan 29. PMID 30824209
- [Background] Strandell A. The influence of hydrosalpinx on IVF and embryo transfer: a review. Hum Reprod Update. 2000 Jul-Aug;6(4):387-95. doi: 10.1093/humupd/6.4.387. PMID 10972525
- [Background] Tsiami A, Chaimani A, Mavridis D, Siskou M, Assimakopoulos E, Sotiriadis A. Surgical treatment for hydrosalpinx prior to in-vitro fertilization embryo transfer: a network meta-analysis. Ultrasound Obstet Gynecol. 2016 Oct;48(4):434-445. doi: 10.1002/uog.15900. Epub 2016 Sep 13. PMID 26922863